CLINICAL TRIAL: NCT00680173
Title: Analysis of Gene Expression of PBMC in the Hepatitis C Virus Genotype 1b-infected Patients During Peg-interferon-α Plus Ribavirin Combination Therapy
Brief Title: Peripheral Blood Mononuclear Cell (PBMC) Gene Expression in HCV Genotype 1 Patients
Acronym: PBMC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wan-Long Chuang, M.D., PhD., Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KMUH-IRB- 950419
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Single nucleotide polymorphisms; Sustained virological response; Peginterferon; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 15 patients with HCV genotype 1 infection receiving peginterferon plus ribavirin achieve a sustained virological response
  Interventions: Drug: pegylated interferon alpha 2a and plus ribavirin
- B (Active Comparator): 15 patients with HCV genotype 1 infection receiving peginterferon plus ribavirin did not achieve a sustained virological response
  Interventions: Drug: pegylated interferon alpha 2a and plus ribavirin

INTERVENTIONS:
Drug: pegylated interferon alpha 2a and plus ribavirin — pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 24 weeks, follow up for 24 weeks
  Other Names: PEGASYS®

SUMMARY:
Our previous collaborative studies has developed a molecular diagnosis tool, which is characterized with a prediction model consisting single nucleotide polymorphisms (SNPs), for assessing the efficacy of interferon combined therapy for chronic hepatitis C (CHC) patients prior to treatment.

Aims of this project:

1. To analyze and validate the gene expression profiling dependent of treatment response to peg-interferon-α plus ribavirin combination therapy in CHC genotype-1 patients.
2. To select the candidate genes and establish a monitoring model assessing the efficacy of interferon treatment.

DETAILED DESCRIPTION:
A combination of pegylated-interferon (PEG-IFN) with ribavirin has been the choice for treating chronic hepatitis C (CHC) patients. In addition to the high cost, the treatment takes 6 to 12 months and often brings significant adverse reactions to some patients. It would therefore be beneficial to include a pre-treatment evaluation and post-treatment monitoring system to maximize the efficacy of CHC therapy. We have established a molecular diagnosis tool for assessing the efficacy of interferon combined therapy for CHC patients prior to treatment. This diagnostic tool is characterized with a prediction model consisting single nucleotide polymorphisms (SNPs) strongly associated with interferon efficacy in treating CHC patients. The prediction model has been validated by hepatitis C samples in Taiwan, and it achieved 80 % accuracy, higher than the current efficacy rates. Supplemented with the viral genotype information would further increase the prediction accuracy to 85%.

In this project, we aim to analyze patients' gene expression profiling during the treatment. The current study will focus on 30 PEG-IFN and ribavirin treated patients with HCV genotype 1 infection. After the responding status of those patients has been confirmed, we will compare gene expression profiling among the different responses before and during treatment. By using this information, we can properly select the candidate genes, and establish a monitoring model with these biomarkers. This monitoring model can thus be applied to assess the efficacy of PEG-IFN plus ribavirin combination treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >18 years of age
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA
* Liver biopsy findings consistent with the diagnosis of chronic hepatitis C infection with or without compensated cirrhosis (Exception: hemophiliacs in whom biopsy is medically contra-indicated do not require biopsy.)
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Present therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* Co-infection with active hepatitis A, hepatitis B and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Clinical evidence of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption>40 g/day) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hgb <11 g/dL in women or <12 g/dL in men at screening
* Any patient with major thalassemia
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated
* Evidence or history of hepatocellular carcinoma
* Local or Systemic malignancy unstable status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Efficacy - Sustained virological response (SVR), HCV RNA seronegative by PCR throughout 24-week off-treatment period. | 1.5 year

SECONDARY OUTCOMES:
Rapid virologic response (RVR), HCV RNA seronegative by PCR at week 4. | 1.5 year
Early virological response (EVR), by PCR-negative or at least 2 logs decline from baseline of serum HCV RNA at 12 weeks of treatment. | 1.5 year
Safety - adverse event rate and profile | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Long Chuang, MD, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Dai CY, Chuang WL, Hsieh MY, Lee LP, Hou NJ, Chen SC, Lin ZY, Hsieh MY, Wang LY, Tsai JF, Chang WY, Yu ML. Polymorphism of interferon-gamma gene at position +874 and clinical characteristics of chronic hepatitis C. Transl Res. 2006 Sep;148(3):128-33. doi: 10.1016/j.trsl.2006.04.005. PMID 16938650
- [Background] Houldsworth A, Metzner M, Rossol S, Shaw S, Kaminski E, Demaine AG, Cramp ME. Polymorphisms in the IL-12B gene and outcome of HCV infection. J Interferon Cytokine Res. 2005 May;25(5):271-6. doi: 10.1089/jir.2005.25.271. PMID 15871664
- [Background] Naito M, Matsui A, Inao M, Nagoshi S, Nagano M, Ito N, Egashira T, Hashimoto M, Mishiro S, Mochida S, Fujiwara K. SNPs in the promoter region of the osteopontin gene as a marker predicting the efficacy of interferon-based therapies in patients with chronic hepatitis C. J Gastroenterol. 2005 Apr;40(4):381-8. doi: 10.1007/s00535-005-1558-3. PMID 15868370
- [Background] Suzuki F, Arase Y, Suzuki Y, Tsubota A, Akuta N, Hosaka T, Someya T, Kobayashi M, Saitoh S, Ikeda K, Kobayashi M, Matsuda M, Takagi K, Satoh J, Kumada H. Single nucleotide polymorphism of the MxA gene promoter influences the response to interferon monotherapy in patients with hepatitis C viral infection. J Viral Hepat. 2004 May;11(3):271-6. doi: 10.1111/j.1365-2893.2004.00509.x. PMID 15117331